CLINICAL TRIAL: NCT00006453
Title: A Randomized Phase III Study Comparing Gemcitabine Plus Carboplatin Versus Carboplatin Monotherapy in Patients With Advanced Epithelial Ovarian Carcinoma Who Failed First-Line Platinum-Based Therapy
Brief Title: Carboplatin With or Without Gemcitabine in Treating Patients With Advanced Ovarian Epithelial Cancer That Has Not Responded to Previous Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AGO Study Group (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067993; AGOSG-OVAR-2.5; CAN-NCIC-OV15; EORTC-55005; EU-20064; NCI-V00-1601
Record Dates: First submitted 2000-11-06; First posted 2003-07-28 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known if carboplatin is more effective with or without gemcitabine for ovarian epithelial cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of carboplatin with or without gemcitabine in treating patients who have advanced ovarian epithelial cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare time to progression in patients with advanced ovarian epithelial carcinoma who failed prior first-line platinum-based therapy when treated with carboplatin with or without gemcitabine.
* Compare response rate, duration of response, and survival time of patients treated with these regimens.
* Compare the toxicity of these treatment regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to progression-free time (6-12 months vs more than 12 months), type of prior first-line therapy, and bidimensionally measurable disease (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive carboplatin IV over 30-60 minutes on day 1 and gemcitabine IV over 30-60 minutes on days 1 and 8.
* Arm II: Patients receive carboplatin IV as in arm I. Treatment in both arms repeats every 3 weeks for up to 6-8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, before each subsequent chemotherapy course, and at 50 days after study.

Patients are followed at 50 days, every 2 months for 1 year, and then every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 350 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial carcinoma not amenable to curative surgery or radiotherapy

  * Evidence of recurrence or progression 6 months after discontinuation of prior first-line platinum-containing regimen
* No tumor of borderline malignancy
* Evaluable disease outside previously irradiated area
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Not specified

Renal:

* Glomerular filtration rate greater than 50 mL/min

Other:

* No concurrent active infection
* No other primary malignancy except carcinoma in situ of the cervix or adequately treated basal cell skin cancer
* No other concurrent serious systemic disorder

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 1 prior platinum-based chemotherapy regimen
* No prior gemcitabine
* No other concurrent cytotoxic or antineoplastic treatment

Endocrine therapy:

* At least 3 weeks since prior hormonal therapy
* Concurrent hormone replacement therapy allowed
* Concurrent steroid antiemetics allowed

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy (limited to the small pelvis)
* Concurrent palliative radiotherapy to nontarget lesions allowed

Surgery:

* See Disease Characteristics

Other:

* At least 3 weeks since other prior investigational agents

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobus Pfisterer, MD, Study Chair — University Hospital Schleswig-Holstein; Angel J. Lacave, MD, PhD, Study Chair — Hospital Universitario Central de Asturias; Marie Plante, MD, Study Chair — Centre Hospitalier Universitaire de Quebec
Locations (74):
- St. Mary's/Duluth Clinic Health System, Duluth, Minnesota, United States
- Canada (73):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Lethbridge Cancer Clinic, Lethbridge, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Nanaimo Cancer Clinic, Nanaimo, British Columbia
  - Penticton Regional Hospital, Penticton, British Columbia
  - British Columbia Cancer Agency - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - St. Paul's Hospital - Vancouver, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Cancer Centre, Victoria, British Columbia
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Doctor Leon Richard Oncology Centre, Moncton, New Brunswick
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cape Breton Cancer Centre, Sydney, Nova Scotia
  - Royal Victoria Hospital, Barrie, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Hamilton and Disrict Urology Association, Hamilton, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Grand River Regional Cancer Centre, Kitchner, Ontario
  - London Health Sciences Centre, London, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - Trillium Health Centre, Mississauga, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - York County Hospital, Newmarket, Ontario
  - North York General Hospital, Ontario, North York, Ontario
  - Male Health Centre/CMX Research Inc., Oakville, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Oncology Clinic, Peterborough, Ontario
  - Algoma District Medical Group, Sault Ste. Marie, Ontario
  - Scarborough Hospital - General Site, Scarborough Village, Ontario
  - Hotel Dieu Health Sciences Hospital - Niagara, St. Catharines, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Mount Sinai Hospital - Toronto, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Women's College Campus, Sunnybrook and Women's College Health Science Center, Toronto, Ontario
  - Saint Joseph's Health Centre - Toronto, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Cancer Care Ontario - Windsor Regional Cancer Centre, Windsor, Ontario
  - Queen Elizabeth Hospital, PEI, Charlottetown, Prince Edward Island
  - Complexe Hospitalier de la Sagamie, Chicoutimi, Quebec
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Centre Hospitalier Regional de Lanaudiere, Joliette, Quebec
  - L'Hotel Dieu de Levis, Lévis, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier de l'Universite' de Montreal, Montreal, Quebec
  - Hotel Dieu de Montreal, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Hopital Du Sacre-Coeur de Montreal, Montreal, Quebec
  - Kells Medical Research Group Inc., Pointe-Claire, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - Centre Hospitalier Regional de Rimouski, Rimouski, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
  - Lions Gate Hospital, North Vancouver
  - Toronto Urology Study Group, Toronto

REFERENCES:
- [Result] Pfisterer J, Plante M, Vergote I, et al.: Gemcitabine/carboplatin (GC) vs. carboplatin (C) in platinum sensitive recurrent ovarian cancer (OVCA). Results of a Gynecologic Cancer Intergroup randomized phase III trial of the AGO OVAR, the NCIC CTG and the EORTC GCG. [Abstract] J Clin Oncol 22 (14 Suppl): A-5005, 450s, 2004.
- [Result] Pfisterer J, Vergote I, Du Bois A, Eisenhauer E; AGO-OVAR,; NCIC CTG; EORTC GCG. Combination therapy with gemcitabine and carboplatin in recurrent ovarian cancer. Int J Gynecol Cancer. 2005 May-Jun;15 Suppl 1:36-41. doi: 10.1111/j.1525-1438.2005.15355.x. PMID 15839957
- [Result] Vergote I, Plante M, Richter B, et al.: Improved progression free survival (PFS) and quality of life (QOL) in a randomised study comparing gemcitabine/carboplatinum (GC) vs. carboplatin (C) in platinum sensitive ovarian cancer (OVCA). [Abstract] Int J Gynecol Cancer 14 (Suppl 1): A-155, 45, 2004.
- [Result] Kurzeder C, Zhao L, Eisenhauer EA, et al.: The impact of dose intensity on the efficacy of gemcitabine plus carboplatin (GC) therapy for recurrent platinum-sensitive ovarian cancer (PSOC): A retrospective analysis of AGO-OVAR 2.5. [Abstract] J Clin Oncol 29 (Suppl 15): A-5088, 2011.
- [Result] Pfisterer J, Plante M, Vergote I, du Bois A, Hirte H, Lacave AJ, Wagner U, Stahle A, Stuart G, Kimmig R, Olbricht S, Le T, Emerich J, Kuhn W, Bentley J, Jackisch C, Luck HJ, Rochon J, Zimmermann AH, Eisenhauer E; AGO-OVAR; NCIC CTG; EORTC GCG. Gemcitabine plus carboplatin compared with carboplatin in patients with platinum-sensitive recurrent ovarian cancer: an intergroup trial of the AGO-OVAR, the NCIC CTG, and the EORTC GCG. J Clin Oncol. 2006 Oct 10;24(29):4699-707. doi: 10.1200/JCO.2006.06.0913. Epub 2006 Sep 11. PMID 16966687